CLINICAL TRIAL: NCT04306107
Title: Prone Position in Non-Invasive Ventilation and High-Flow Oxygen Therapy
Acronym: ProPNIVFlow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Morales Meseguer (Other)
Responsible Party: Principal Investigator, Miguel Filipe Martins de Matos Navarro Guia, MD, Hospital General Universitario Morales Meseguer
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-03-2020; 10-03-2020 2 (Other: International Association Noninvasive Ventilation)
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Evaluation of Prone Position Effect During NIV and HFNC on Acute Hypoxemic Respiratory Failure
Keywords: Noninvasive ventilation; High-flow nasal oxygen therapy; Prone position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NIV with prone position (Experimental): Use of prone position during NIV
  Interventions: Device: Prone position during non-invasive respiratory support
- NIV (conventional) (Placebo Comparator): NIV on conventional position
  Interventions: Device: Prone position during non-invasive respiratory support
- HFNC on prone position (Experimental): Prone position during HFNC
  Interventions: Device: Prone position during non-invasive respiratory support
- HFNC (conventional) (Placebo Comparator): HFNC on conventional position
  Interventions: Device: Prone position during non-invasive respiratory support

INTERVENTIONS:
Device: Prone position during non-invasive respiratory support — HFNC and NIV application with patient on prone position
  Other Names: HFNC and NIV application with patient on prone position

SUMMARY:
The aim of this trial is to study the effect of prone position during NIV and HFNC on acute hypoxemic respiratory patients.

DETAILED DESCRIPTION:
Inclusion Criteria:

Adult patients with:

• ARDS/pneumonia/acute hypoxemic respiratory failure with PaO2/FiO2 between 150 and 300 (on 5 cmH2O PEEP level)

Exclusion Criteria

* General NIV or HFNC contraindications
* Immediate need for IOT
* Prone position intolerance
* Patients refusal to participate

Interventions:

* Prone position for 2-4 hours twice a day, for 3 days (first 3 days since admission to ICU)
* Nurse surveilance: at least every 15 minutes

Outcomes:

* Need for IOT
* Effects on the measurements specified above (particularly PaO2/FiO2)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with:

  * ARDS/pneumonia/acute hypoxemic respiratory failure with PaO2/FiO2 between 150 and 300 (on 5 cmH2O PEEP level)

Exclusion Criteria:

* General NIV or HFNC contraindications
* Immediate need for IOT
* Prone position intolerance
* Patients refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Oro-tracheal entubation | 1 month
  Oro-tracheal entubation avoidance

SECONDARY OUTCOMES:
PaO2/FiO2 | 1 month
  Effect of prone position on PaO2/FiO2

IPD SHARING:
Plan to Share IPD: Undecided